CLINICAL TRIAL: NCT03628404
Title: Defining the Genetic Etiology of Alzheimer's Disease in the Faroe Islands
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faroese Hospital System (Other)
Responsible Party: Principal Investigator, Maria Skaalum Petersen, Associate professor, Faroese Hospital System
Other Study IDs: AD
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer disease; Dementia; Faroe Islands; Isolated population; Environmental exposure
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma and buffy coat
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators established the Faroese Alzheimer's Cohort with the aim to unravel genetic and environmental factors that influence the risk and/or susceptibility of Alzheimers disease (AD). It is believed the Faroese population represents a unique opportunity due to its characteristics as a geographic, environmental and genetic isolate with a homogeneous genetic background and founder effects. It has an 'engaged' population with superbly detailed genealogy going 400 years back, unfettered patient access to health care, traditionally high participation rates in research and low probability of losing subjects to follow-up, and presents a unique opportunity to more readily identify genetic and environmental factors involved in AD.

The specific aims of this project are:

1. Enrolment of patients with AD, incl.1st degree family members of selected familial patients and age and gender matched control subjects.
2. Detailed genealogical investigation of patients with Alzheimer's disease
3. Identify genes influencing risk and/or susceptibility of AD in the Faroese population

DETAILED DESCRIPTION:
The aim of the study is to unravel genetic and environmental factors that influence the risk and/or susceptibility of AD. Thus, subjects with AD and family members when there is a strong history of AD are being recruited. Data collection includes a blood sample, clinical phenotype data from hospital records, standardized assessment scales (e.g. Geriatric Depression Scale (GDS), Neuropsychiatric Inventory Questionnaire (NPI-Q), Functional Activities Questionnaire (FAQ-IADL), tests of mental function (Mini Mental State Examination (MMSE) and Addenbrooke's Cognitive Examination (ACE)) and family and lifestyle/environmental questionnaire. Furthermore are control subjects being recruited where data includes a blood sample, MMSE and a lifestyle/environmental questionnaire.

Initial genetic analyses will focus on known genetic risk factors for AD by looking at the most highly associated single nucleotide polymorphisms in loci harboring e.g. apolipoprotein E (APOE)/Translocase Of Outer Mitochondrial Membrane 40 (TOMM40), MAPT, Phosphatidylinositol Binding Clathrin Assembly Protein (PICALM). Subsequent analyses will focus on genome-wide array genotyping of ~ 1.8 million markers, e.g. to accommodate the population structure. Finally, patients with a family history of AD who cannot be explained by the before mentioned analysis will be subject to exome sequencing. Exposure analyses will focus on persistant organic pollutants, e.g. polychlorinated biphenyls (PCBs), perfluorinated alkylated substances (PFAS) and also mercury.

The investigators believe the Faroese population presents a unique opportunity to more readily identify genetic and environmental factors involved in AD due to its characteristics as a geographic, environmental and genetic isolate with a homogeneous genetic background.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia (cases)
* Age and gender matched to cases (controls)
* Close relatives to an individual with dementia (family members)

Exclusion Criteria:

* No exclusion criteria (cases and family members)
* Sign of dementia assessed by MMSE (controls)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a population based study conducted in the Faroe Islands, a small island population with approximately 50.000 inhabitants. Individuals diagnosed with dementia are being recruited from the only Dementia Clinic on the islands. Family members are also recruited. Control subjects are randomly selected from the Faroese Population Registry, matched by sex and age to the cases. Te
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sequenom iPLEX genotyping and exome sequencing to identify and characterize genetic contributions to etiology of Alzheimer disease and other dementias | At baseline
  Genetic cause of disease

SECONDARY OUTCOMES:
Influence of polychlorinated biphenyl exposure on the risk of AD | At baseline
  Polychlorinated biphenyls levels measured in serum
Influence of perfluorinated alkylated substance exposure on the risk of AD | At baseline
  Perfluorinated alkylated substances (PFAS) levels measured in serum
Influence of mercury exposure on the risk of AD | At baseline
  Mercury levels measured in blood
MMSE | At baseline
  Mini Mental State Examination
ACE | At baseline
  Addenbrooke's cognitive examination
NPI-Q | At baseline
  The Neuropsychiatric Inventory
FAQ IADL | At baseline
  Functional Activities Questionnaire / Functional Assessment Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Faroses Hospital System, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: Undecided